CLINICAL TRIAL: NCT01046968
Title: The Use of LeptiCore® in Reducing Fat Gain and Managing Weight Loss in Patients With Metabolic Syndrome
Brief Title: Lepticore in Metabolic Syndrome and Weight Loss
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Yaounde 1 (Other)
Collaborators: Cameroon Nutritional Science Society (Unknown)
Responsible Party: Pr. Julius Oben - Head of Laboratory of Nutrition & Nutritional Biochemistry, University of Yaounde 1
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LNNB232
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-07

CONDITIONS: Obesity; Hyperlipidemia; Hyperglycemia
Keywords: Obesity; metabolic syndrome; C-reactive protein; Leptin
MeSH Terms: conditions — Obesity; Hyperlipidemias; Hyperglycemia; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lepticore (Experimental)
  Interventions: Dietary Supplement: Lepticore

INTERVENTIONS:
Dietary Supplement: Lepticore — 300 mg twice daily
  Other Names: Plant based polysaccharides

SUMMARY:
Metabolic syndrome is directly related to obesity. This study investigated the use of a plant based formulation to improve on the condition of people with metabolic syndrome.

DETAILED DESCRIPTION:
LeptiCore is a proprietary combination of various ingredients which have been shown to have properties which could be beneficial to weight loss in obese and overweight human subjects. This study evaluates the effect of Lepticore on bodyweight as well as parameters associated with obesity and metabolic syndrome.

The study was an 8 week randomized, double-blind, placebo-controlled design involving 92 obese (mean BMI>30kg/m2) participants (37 males; 55 females; ages 19-52; mean age = 30.7). The participants were randomly divided into three groups: placebo (n=30), LeptiCore formula A (low dose) (n=31) and LeptiCore formula B (high dose) (n=31). Capsules containing the placebo or active formulations were administered twice daily before meals with 300 ml of water. None of the participants followed any specific diet nor took any weight-reducing medications for the duration of the study. A total of 12 anthropomorphic and serological measurements were taken at the beginning of the study and after 2, 4, 6, and 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30 kg/m2
* Total cholesterol >200 mg/dl
* LDL cholesterol >160 mg/dl
* HDL cholesterol <40 mg/dl; triglycerides >150 mg/dl
* Fasting blood glucose >100 mg/dl
* Blood pressure >130/85 mmHg.

Exclusion Criteria:

* Morbid obesity (BMI >40 kg/m2 )
* Diabetes mellitus requiring daily insulin management
* Pregnancy/lactation
* Active infection
* Systemic disease such as HIV/AIDS,
* Use of any cholesterol-lowering medications 30 days prior to study
* Enrollment in another clinical study within the past 6 months.

Ages: 19 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Improvement of symptoms of metabolic syndrome | 8 weeks

SECONDARY OUTCOMES:
Change in weight | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julius E Oben, PhD, Principal Investigator — University of Yaounde 1
Locations (1):
- Laboratory of Nutrition and Nutritional Biochemistry, Yaoundé, Centre Region, Cameroon